CLINICAL TRIAL: NCT02858219
Title: A Pilot Study of the Effects of Botulinum Toxin in the Treatment of Provoked Vestibulodynia
Acronym: VESTIBULE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: API/2011/20
Record Dates: First submitted 2016-08-01; First posted 2016-08-08 (Estimated); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Vestibulodynia
Keywords: Botulinum toxin; Pain improvement
MeSH Terms: conditions — Vulvodynia | interventions — Botulinum Toxins, Type A; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Botulinum toxin (Experimental): Injection of 50 units (50U) botulinum toxin type A (powder), reconstituted in 1 mL physiologic saline solution in each perineal muscle (100 units in total).
  First injection at day 1 and. A second injection is scheduled at 3 months, only if there is a 50% or more pain improvement compared to baseline (pain measured with Visual Analogic Scale).
  Interventions: Drug: Botulinum Toxin Type A; Other: Indexes
- Saline solution (Placebo Comparator): Injection of 1 mL physiologic saline solution in each perineal muscle. A second injection is scheduled at 3 months, only if there is a 50% or more pain improvement compared to baseline (pain measured with Visual Analogic Scale).
  Interventions: Other: Saline solution; Other: Indexes

INTERVENTIONS:
Drug: Botulinum Toxin Type A
  Arms: Botulinum toxin
Other: Saline solution
  Arms: Saline solution
Other: Indexes — Visual Analogic Scale (VAS), Female Sexual Function Index (FSFI), Dermatology Life Quality Index (DLQI)

SUMMARY:
The main objective of this study is to compare the efficacy of botulinum toxin injections on vestibulodynia pain compared to a group treated with a placebo.

ELIGIBILITY:
Inclusion Criteria:

* Subject refractory to conventional treatments (tricyclic antidepressants and benzodiazepines at analgesic doses, biofeedback physical therapy)
* Negative screening test results
* Notified associated factors
* Menopause, surgically sterilized women or women using effective contraceptive method
* Good understanding and predictable adherence to the protocol
* beneficiary/affiliated to French social security/social healthcare
* signed Informed Consent Form

Exclusion Criteria:

* Predictable poor adherence
* Pregnant or breastfeeding women
* Myasthenia
* Treatment with aminoglycosides
* Major mental disorders
* Underlying etiology
* Vulnerable subjects (particularly adults under guardianship)
* Any reason deemed relevant by the investigator
* Current or former (in the last 3 months) participation to another clinical trial

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2010-05-04 (Actual); Primary Completion 2019-02-11 (Actual); Study Completion 2019-02-11 (Actual)

PRIMARY OUTCOMES:
Pain improvement | 3 months
  Significant improvement of pain on contact in the treated group, compared to placebo group, measured with Visual Analogic Scale

CONTACTS AND LOCATIONS:
Overall Officials: Fabien Pelletier, MD, Principal Investigator — Centre Hospitalier Universitaire de Besancon
Locations (2):
- France (2):
  - CHU Besançon, Besançon
  - Hôpital Tenon, Paris

IPD SHARING:
Plan to Share IPD: No